CLINICAL TRIAL: NCT03084094
Title: Transcranial Direct Current Stimulation and Its Therapeutic Potentiality in Different Populations
Brief Title: Neuromodulation and Its Therapeutic Potentiality in Different Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Karime Andrade Mescouto, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS in fibromyalgia
Record Dates: First submitted 2017-03-07; First posted 2017-03-20 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; tDCS
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M1 (Experimental): Transcranial direct current Stimulation in primary motor cortex
  Interventions: Device: Transcranial Direct Current Stimulation
- DLPFC (Experimental): Transcranial direct current Stimulation in the dorsolateral pre-frontal cortex
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham (Sham Comparator): sham stimulation
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Non invasive brain modulation at a 2mA current during 20minutes

SUMMARY:
One of the big challenges faced by researchers who act in rehabilitation science is the capacity to dispose integrative approaches for its utilization in clinical practice. The border profile of a physiotherapy researcher is to be in front of applied research amplification in experimental integrative approaches, involving the study of behavioral and physiological variables.

The rehabilitation process transcends the systems physiology and encompasses the cognitive behavioral feature of being adapted to the environment that surround us. It is now known by the scientific rehabilitation community the necessity for evidence based therapies and even more, therapeutic innovation. In both conditions, of health and illness, various options to use integrative approaches are today available in physiotherapy, including behavioral and physiological profiles of the individuals during physical activities, response to stress and in the field of chronic pain.

It is in the clinical routine of numerous rehabilitation centers the treatment of diseases that causes pain, being the leading figure in a physiotherapist work process. The innovative study of resources that can alter the pain state of this patients becomes primordial for routine clinical use, low cost and easy to apply. The therapeutic treatment for pain offered by a physiotherapist need new investigative options based in evidences from the association between the neuronal, behavioral and physiological responses where the brain is the central organ of this regulation. In this context, become increasingly more necessary the construction of investigative approaches in the purpose of reaching the clinical practice, in a reduced time lapse, once the great volume of information produced globally does not impact in short or medium term in new therapeutic recommendations.

Among the various chronic painful entities, it is presented the fibromyalgia (FM), painful diabetic polyneuropathy and primary dysmenorrhea because of its painful pathogenic complexity and its limited therapeutic against pain in rehabilitation process. The 3 painful entities presents the central nervous system as main participant of neurogenesis and maintenance of the painful state.

It is primordial importance that rehabilitation science improve methods of non invasive brain neuromodulation that allows, through excitation or inhibition of specific cortical areas in order to produce pain inhibition, providing a simple and low cost treatment to clinical routine. Technological advances and non invasive techniques to modulate brain function has been developed, among which transcranial direct current stimulation (tDCS) stands out. Basically, electrodes are placed in targeted brain regions that you want to stimulate or inhibit. Posteriorly, is applied a continuous electric current (0,4 - 2 mA) for a 3-20 minutes period, in order to modify cortical excitability. The stimulus of the anodic current increases cortical excitability whereas the stimulus of the cathodic current has an inhibitory effect.

Few are the research groups that address the issue of fibromyalgia, painful diabetic polyneuropathy and primary dysmenorrhea and the application of tDCS as research focus, being a border area for rehabilitation science and great potential in clinical use. Preliminary studies associates the use of tDCS with the decrease of painful state, however an approach of physical function and behavioral results needs greater investigation.

The purpose of the presented project is to present the tDCS as a new modality in physical rehabilitation for the patient with chronic pain of the 3 entities mentioned above. The study proposal is to present behavioral, social and physical results of tDCS application in this patients, suggesting a better quality of life and functionality of the individual.

ELIGIBILITY:
Inclusion Criteria:

- Female gender aged from 18 to 65 year old, having a clinical diagnosis of Fibromyalgia given by a rheumatologist.

Exclusion Criteria:

* Non-regulated psychiatric disorders (bipolar, main depression, schizophrenia)
* Performing other types of treatment during the research
* Performing physical activities

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain at 2 weeks | 1 week prior to treatment (Baseline) and 1 week during treatment
  Diary of Pain
Change from Baseline Pain at 5 weeks | 1 week prior to treatment, day 1 of treatment, last day of treatment (day 5), 7 days, 14 days and 21 days after treatment
  Pressure Pain Threshold and Tolerance by an algometer
Change from Baseline Pain at 5 weeks | 1 week prior to treatment, day 1 of treatment, last day of treatment (day 5), 7 days, 14 days and 21 days after treatment
  Visual Analogue Scale

SECONDARY OUTCOMES:
Functional Capacity | 1 week prior to treatment, last day of treatment (day 5),7 days, 14 days and 21 days after treatment
  Fibromyalgia Impact Questionnaire
Mood | 1 week prior to treatment, last day of treatment (day 5),7 days, 14 days and 21 days after treatment
  Beck Depression Inventory
Anxiety | 1 week prior to treatment, last day of treatment (day 5),7 days, 14 days and 21 days after treatment
  Hamilton Anxiety Scale
Positive and negative affect | 1 week prior to treatment, last day of treatment (day 5),7 days, 14 days and 21 days after treatment
  Positive and Negative Affect Schedule

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Onofre Lopes, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No